CLINICAL TRIAL: NCT01713920
Title: Efficacy and Tolerability of Combination Antihypertensive Drug in Non-Responders to Angiotensin Receptor Blocker(ARB) monoTHerapy Using 24h ABPM.
Brief Title: Efficacy and Tolerability of Combination Antihypertensive Drug in Non-Responders to ARB monoTHerapy Using 24h ABPM
Acronym: EARTH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sang Hyun Ihm, MD PhD (Other)
Collaborators: Daiichi Sankyo Korea Co., Ltd. (Industry); Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor-Investigator, Sang Hyun Ihm, MD PhD, Associate Professor , Division of Cardiology, Department of Internal Medicine, The Catholic University of Korea
Organization: The Catholic University of Korea (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EARTH
Record Dates: First submitted 2012-10-22; First posted 2012-10-25 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SEVIKAR (Experimental): Subjects who are eligible for the inclusion and exclusion criteria will be treated with Sevikar 5/20mg for 4 weeks. If subjects fail to reach the SBP threshold of SeSBP≥ 140mmHg after 4-week treatment, they will receive Sevikar 5/40mg for 4 weeks. At the end of 4-week treatment, subjects who fail to reach SBP threshold will receive Sevikar 10/40mg for 4 weeks. Subjects who can reach SBP threshold will continue to treat with current dose until 12 weeks.
  Interventions: Drug: SEVIKAR

INTERVENTIONS:
Drug: SEVIKAR
  Other Names: amlodipine + olemsartan

SUMMARY:
A majority of Korean doctors tend to add other antihypertensive rather than to titrate the same drug.

However, we try to induce doctors to titrate the Sevikar than to add other antihypertensive if patients are not controlled with Sevikar 5/20mg(amlodipine 5mg + omlesartan 20mg). As above, for patients who are not controlled with Sevikar 5/20mg, doctors will proceed to other prescription pattern with other choices of titration to Sevikar 5/40, 10/40mg.

It is important to evaluate BP lowering efficacy of Sevikar through the titration step in patients uncontrolled with Sevikar low dose. Thus, this study is designed to demonstrate the efficacy of Sevikar by titration in patients who are not controlled their BP with low dose of Sevikar.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects > 55 years
2. Subject who has consent to participate by signing on the informed consent form
3. Uncontrolled hypertensive patients defined as:

   * Uncontrolled hypertensive: subjects who are mean SBP ≥ 140 mmHg after being treated with ARB(Valsartan 80mg or Candesartan 8mg) monotherapy during at least 4 weeks.

Exclusion Criteria:

1. Secondary hypertension
2. SeSBP ≥ 180mmHg
3. SeSBP difference ≥ 20mmHg or SeDBP difference ≥ 10mmHg
4. A history of hypertensive encephalopathy, unstable angina, transient ischemic attack, MI, or any type of revascularization procedure within the last 6 months
5. Heart failure, second- or third-degree heart block, significant arrhythmia or valvular heart disease
6. Significant cardiovascular, cerebrovascular, renal, gastrointestinal, or hematologic disease, at the discretion of investigator
7. Creatinine clearance<20mL/min and Renal artery stenosis, Renal Transplantation, Patients with only one kidney
8. Evidence of liver disease as indicated by alanine transaminase (ALT) and aspartate transaminase (AST) and/or total bilirubin ≥ 3 × the upper limit of normal (ULN)
9. Hyperkalemia (>5.5mmol/L)
10. Patients with sodium depletion is not correct or Patients with fluid depletion is not correct
11. Chronic inflammation
12. Patients with severe eye-related disorders (Retinal bleeding within 6 months, Blindness, Hypertension complications with Retinal micro-aneurysms)
13. Diabetes mellitus
14. Hematologic/oncologic, neurologic and psychiatric diseases
15. Females who were pregnant, breastfeeding, planning a pregnancy or who were of childbearing potential
16. Contraindications for amlodipine, losartan, olmesartan medoxomil, or other ARBs
17. With known allergic reaction, lack of response or contraindication to Angiotensin II receptor antagonists
18. Mean DBP > 110 mmHg
19. Patients who took antihyperlipidemic agents within 30 days
20. Subject who have participated in other clinical trial within the last one month
21. Any subjects who are unable to cooperate with protocol requirements and follow-up procedures or who are in medical condition that is not eligible to be entered in investigators' discretion

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
change in mean 24-hour ABPM SBP | from baseline to Week 12

SECONDARY OUTCOMES:
value of cuff SeSBP/SeDBP | baseline, week 4, week 8 and week 12
change in aortic PWV | from baseline to week 4, week 8, week 12
change in 24-hour ABPM DBP | baseline to week 12
change in hsCRP, HOMA-IR, MAU, Uric acid | from baseline to week 12

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - The Catholic University of Korea Bucheon St. Mary's Hospital, Bucheon-si
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul

REFERENCES:
- [Background] Korean National Health & Nutrition Examination Surveys. Available from: URL://http://knhanes.cdc.go.kr/
- [Background] Hansson L, Zanchetti A, Carruthers SG, Dahlof B, Elmfeldt D, Julius S, Menard J, Rahn KH, Wedel H, Westerling S. Effects of intensive blood-pressure lowering and low-dose aspirin in patients with hypertension: principal results of the Hypertension Optimal Treatment (HOT) randomised trial. HOT Study Group. Lancet. 1998 Jun 13;351(9118):1755-62. doi: 10.1016/s0140-6736(98)04311-6. PMID 9635947
- [Background] ALLHAT Officers and Coordinators for the ALLHAT Collaborative Research Group. The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. Major outcomes in moderately hypercholesterolemic, hypertensive patients randomized to pravastatin vs usual care: The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT-LLT). JAMA. 2002 Dec 18;288(23):2998-3007. doi: 10.1001/jama.288.23.2998. PMID 12479764
- [Background] Dahlof B, Sever PS, Poulter NR, Wedel H, Beevers DG, Caulfield M, Collins R, Kjeldsen SE, Kristinsson A, McInnes GT, Mehlsen J, Nieminen M, O'Brien E, Ostergren J; ASCOT Investigators. Prevention of cardiovascular events with an antihypertensive regimen of amlodipine adding perindopril as required versus atenolol adding bendroflumethiazide as required, in the Anglo-Scandinavian Cardiac Outcomes Trial-Blood Pressure Lowering Arm (ASCOT-BPLA): a multicentre randomised controlled trial. Lancet. 2005 Sep 10-16;366(9489):895-906. doi: 10.1016/S0140-6736(05)67185-1. PMID 16154016
- [Background] Poulter NR, Wedel H, Dahlof B, Sever PS, Beevers DG, Caulfield M, Kjeldsen SE, Kristinsson A, McInnes GT, Mehlsen J, Nieminen M, O'Brien E, Ostergren J, Pocock S; ASCOT Investigators. Role of blood pressure and other variables in the differential cardiovascular event rates noted in the Anglo-Scandinavian Cardiac Outcomes Trial-Blood Pressure Lowering Arm (ASCOT-BPLA). Lancet. 2005 Sep 10-16;366(9489):907-13. doi: 10.1016/S0140-6736(05)67186-3. PMID 16154017
- [Background] Chrysant SG, Melino M, Karki S, Lee J, Heyrman R. The combination of olmesartan medoxomil and amlodipine besylate in controlling high blood pressure: COACH, a randomized, double-blind, placebo-controlled, 8-week factorial efficacy and safety study. Clin Ther. 2008 Apr;30(4):587-604. doi: 10.1016/j.clinthera.2008.04.002. PMID 18498909
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] Mancia G, De Backer G, Dominiczak A, Cifkova R, Fagard R, Germano G, Grassi G, Heagerty AM, Kjeldsen SE, Laurent S, Narkiewicz K, Ruilope L, Rynkiewicz A, Schmieder RE, Boudier HA, Zanchetti A, Vahanian A, Camm J, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Erdine S, Kiowski W, Agabiti-Rosei E, Ambrosioni E, Lindholm LH, Viigimaa M, Adamopoulos S, Agabiti-Rosei E, Ambrosioni E, Bertomeu V, Clement D, Erdine S, Farsang C, Gaita D, Lip G, Mallion JM, Manolis AJ, Nilsson PM, O'Brien E, Ponikowski P, Redon J, Ruschitzka F, Tamargo J, van Zwieten P, Waeber B, Williams B; Management of Arterial Hypertension of the European Society of Hypertension; European Society of Cardiology. 2007 Guidelines for the Management of Arterial Hypertension: The Task Force for the Management of Arterial Hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2007 Jun;25(6):1105-87. doi: 10.1097/HJH.0b013e3281fc975a. No abstract available. PMID 17563527
- [Derived] Chung WB, Ihm SH, Choi YS, Youn HJ. Efficacy of Olmesartan/Amlodipine Single-Pill Combination on 24-h Mean Systolic Blood Pressure Measured by Ambulatory Monitoring in Non-Responders to Valsartan or Candesartan Monotherapy. J Clin Hypertens (Greenwich). 2025 Jan;27(1):e14929. doi: 10.1111/jch.14929. Epub 2024 Nov 6. PMID 39504016